CLINICAL TRIAL: NCT03126292
Title: Promoting Early Child Development in Primary Care for Low-Income Families
Brief Title: Child Development and Primary Care in Low Income Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Reshma Shah, MD, Assistant Professor of Pediatrics, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014-0337_3; K23HD086295 (NIH)
Record Dates: First submitted 2017-04-18; First posted 2017-04-24 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Parenting; Development, Child
Keywords: Medical home; Primary care; Children; Development

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sit Down and Play (Experimental): Families randomized to intervention group will receive Sit Down and Play while they wait in the waiting room to be seen by their primary care provider at current and subsequent well-child visits.
  Interventions: Behavioral: Sit Down and Play
- Handout (Active Comparator): Families in the control group will receive handouts regarding child safety
  Interventions: Other: Child Safety Handout

INTERVENTIONS:
Behavioral: Sit Down and Play — Sit Down and Play (SDP) is designed to be a brief, low-cost intervention that incorporates key theoretical constructs to elicit positive parenting behaviors. It is intended to be delivered by existing clinical staff, nonprofessionals, or volunteers during each of the eight well-child visits between 2-24 months of age while a family waits to be seen by their pediatrician in the examination room.
  Arms: Sit Down and Play
Other: Child Safety Handout — Handout regarding early child safety
  Arms: Handout

SUMMARY:
The objective of this study is to conduct a 12-month pilot longitudinal study of a parent-directed program delivered in a primary care setting serving primarily low-income families. The parent-direction program will be evaluated in a randomized controlled design to determine the feasibility of protocol implementation and to investigate the potential impact on parental outcomes. Process outcomes will include success with recruitment, participant retention, and ability to collect outcome measures. Clinical outcomes will incorporate measures of parental self-efficacy and parenting behaviors, including observational assessments of parent-child interactions.

DETAILED DESCRIPTION:
Enriching parenting behaviors in early childhood promotes child development and offers a promising strategy to reduce future educational disparities. However, current interventions are limited by cost and have not been widely disseminated. Recognized as a target for research to improve early childhood development and subsequent school readiness skills among at-risk families, the primary care setting offers an ideal opportunity to reach the millions of children living in poverty. However, what remains unknown is how to more efficiently leverage the primary care setting to deliver a sustainable and effective preventive program to promote positive parenting behaviors and encourage early childhood development in low-income families. Therefore, the investigators designed Sit Down and Play (SDP) a brief parent-directed program delivered in the primary care setting. Modeled after the widely disseminated literacy program Reach Out and Read and grounded in social cognitive theory, SDP is intended to take place during each pediatric well-child visit occurring in a child's first two years with the goal of promoting positive parenting behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Parent is 18 years or older
* Child is present for a 2 month well-child visit
* Adult present with child at appointment is parent/caregiver of child

Exclusion Criteria:

* Parent is non-English speaking
* Child is acutely sick

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in parental knowledge regarding importance of verbal interactions | 6 and 12 months post-enrollment
  Change in knowledge regarding importance of talking with children less then 2 years of age as measured by the Thirty Million Word Questionnaire
Participation in cognitively stimulating activities | 12 months post enrollment
  Participation in cognitively stimulating activities such as reading and play as measured by the StimQ
Parent-child interactions | 12 months post enrollment
  Observational assessment to assess parental sensitivity, involvement in child activities, and engagement in language experiences utilizing the Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO)

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Shah, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah R, Kennedy S, Clark MD, Bauer SC, Schwartz A. Primary Care-Based Interventions to Promote Positive Parenting Behaviors: A Meta-analysis. Pediatrics. 2016 May;137(5):e20153393. doi: 10.1542/peds.2015-3393. Epub 2016 Apr 19. PMID 27244800
- [Background] Shah RP, Kunnavakkam R, Msall ME. Pediatricians' knowledge, attitudes, and practice patterns regarding special education and individualized education programs. Acad Pediatr. 2013 Sep-Oct;13(5):430-5. doi: 10.1016/j.acap.2013.03.003. Epub 2013 Mar 14. PMID 23707687